CLINICAL TRIAL: NCT02219984
Title: Phase 4 Study on Clinical History of Patients Who Start a Chronic Anticoagulant Treatment
Brief Title: START-Register: Survey on Anticoagulated Patients Register
Status: Recruiting | Type: Observational
Sponsor: GUALTIERO PALARETI (Other)
Collaborators: Arianna Anticoagulazione Foundation (Other)
Responsible Party: Sponsor-Investigator, GUALTIERO PALARETI, Professor in Vascular Medicine, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Organization: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Other Study IDs: 142/2010/O/Oss
Record Dates: First submitted 2014-08-12; First posted 2014-08-19 (Estimated); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Atrial Fibrillation; Venous Thromboembolism; Heart Valve Diseases or Prosthesis
Keywords: Anticoagulation; vitamin K antagonists; Warfarin; low molecular weight heparin; fondaparinux; antithrombotics; Direct oral anticoagulants; dabigatran; rivaroxaban; apixaban; edoxaban; atrial fibrillation; venous thromboembolism
MeSH Terms: conditions — Atrial Fibrillation; Venous Thromboembolism; Heart Valve Diseases | interventions — Anticoagulants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — plasma samples for measurements of anticoagulant drug activity
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- patients anticoagulated
  Interventions: Drug: Anticoagulants

INTERVENTIONS:
Drug: Anticoagulants

SUMMARY:
This is a phase 4 cohort prospective, open, national, multicentre study that collects data on history of patients treated chronically with anticoagulant drugs, including the novel direct oral anticoagulants (DOACs). The Registry is designed solely for observational purposes and is not intended to have any influence on the treatment of the single patients included.

Patients are included when they start the anticoagulant treatment, whatever the drug used, or when they shift from a vitamin K antagonist (VKA) drug to one of the novel direct oral anticoagulants, provided that the therapy is expected to last at least 3 months.

The general aims of the study are to provide a better evaluation of efficacy and safety of different treatment options, and to improve our understanding of the risks/benefits of the various anticoagulant drugs and the different therapy options.

The Registry is open to the participation of clinical centres or individual professionals (now called Participants) that are involved with management of anticoagulated patients.

DETAILED DESCRIPTION:
Participants can include patients with 18 years or more who satisfy the following preset criteria:

* Participants should included patients consecutively to avoid selection bias; criteria to avoid selection bias are proposed to Participants, which should decide the one they want to adopt.
* Patients should have been receiving anticoagulation therapy for no more than 30 days at the time of inclusion, regardless of age, clinical indication for treatment, therapeutic range expected (in cases of treatment with VKAs) and expected duration of the treatment (providing a duration of at least 3 months is foreseen). Patients who have already been receiving chronic anticoagulation therapy for some time may be included if they are switched from VKAs to DOACs or to low molecular weight heparin or to fondaparinux
* Patients not prepared to undergo constant monitoring at their enrolling centres or who take part in phase II or III clinical studies should not be included. Patients who participate in other observational or phase IV studies can be included in the Register.
* All patients must give their informed written consent -- following procedures laid down by local Ethical Committees - for the compilation and conservation on the Register's central database of data regarding their personal clinical histories and anticoagulation treatment patterns and for use of said data.
* All the patients inserted must be followed for at least 1 year, even though an indefinite follow-up of all patients continuing anticoagulation therapy is highly recommended. If in single patients anticoagulation treatment is discontinued within 1 year of inclusion, active participating members should nonetheless keep on compiling (telephonically too) information regarding the possible onset of complications (thrombotic, bleeding clinical events of another nature) till 1 year -follow-up.
* The Participants of the Register must use a computer programme as database - for all the information to be collected. The computer programme must meet the features requested by the Executive Committee of the Registry and must be able to send the information to the centralised database via internet and connection to the web site. By way of alternative the Participants can use the "Simple-START" software provided free by the Registry.
* As criterion for safeguarding the privacy of patients, every patient inserted in the Registry is identified by a "Patient log" which includes the identification code of the enrolling Participant and the identification code of each single patient, using the computer database programme used by the Participant. The enrolling Participant is committed to keeping for the whole duration of the Register the whole demographic data of each patient associated with the Patient log".
* Are excluded patients who: have < 18 years age, are not willing to sign informed consent, are not ready to submit to constant monitoring, participate in phase II or III clinical studies
* Follow-Up All the patients inserted must be followed for at least 1 year even though an indefinite follow up of all patients continuing anticoagulation therapy is strongly recommended. If anticoagulation therapy is interrupted in single patients within 1 year of insertion the Participants must still continue to collect (even telephonically) data regarding the possible onset of complications (thrombotic, bleeding or other clinical events) for 1 year of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* age >= 18 years

Exclusion Criteria:

* < 18 years
* not willing to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Are included in the Registry patients who need chronic anticoagulation for atrial fibrillation, or venous thromboembolism, or heart valve diseases or prosthesis, or other clinical conditions requiring anticoagulation.
  For the sampling method, participants are instructed to choose and declare one modality of inclusion for VKA treated patients: one week per month, or one day per week (always the same), etc. For patients treated with DOACs (low number in our country) it is recommended to include all patients progressively
Sampling Method: Probability Sample
Enrollment: 15410 (Estimated)
Dates: Start 2011-10 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
incidence of complications (number per cent patient-years of treatment) | at 1 year of follow-up
  from date of inclusion in the registry until the date of first documented major complication or date of death from any cause, whichever came first, assessed up to 5 years.

SECONDARY OUTCOMES:
Percentage of Time in the therapeutic range (TTR) | at 1 year
  This only applies to patients who receive VKAs for treatment; from date of inclusion in the registry until the date of VKA treatment was stopped, or date of death from any cause, whichever came first, assessed up to 5 years

OTHER OUTCOMES:
percentage of patients who stop anticoagulant treatment | at 1 year
  This applies only to patients anticoagulated for atrial fibrillation; from date of inclusion in the registry until the date anticoagulant treatment was discontinued, or date of death from any cause, whichever came first, assessed up to 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- S. Orsola-Malpighi University hospital, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Menichelli D, Gazzaniga G, Poli D, Palareti G, Antonucci E, Pani A, Pignatelli P, Pastori D; START2 Register Investigators. Real-world use of direct oral anticoagulants in atrial fibrillation patients with moderate/severe chronic kidney disease: a propensity score matched analysis from the START registry. Clin Res Cardiol. 2025 Nov 3. doi: 10.1007/s00392-025-02765-7. Online ahead of print. PMID 41182346
- [Derived] Menichelli D, Antonucci E, Gazzaniga G, Poli D, Armentaro G, di Carlo G, Marcucci R, Calabro P, Cesaro A, Palareti G, Sciacqua A, Pignatelli P, Pastori D; START 2 Collaborators *. Atrial Fibrillation, Heart Failure Phenotypes, and Mortality Risk in the Nationwide START Registry: A Propensity Score Matching Analysis. J Am Heart Assoc. 2025 Jun 17;14(12):e042586. doi: 10.1161/JAHA.125.042586. Epub 2025 Jun 16. PMID 40519207
- [Derived] Antonucci E, Poli D, Tosetto A, Pengo V, Tripodi A, Magrini N, Marongiu F, Palareti G; START-Register. The Italian START-Register on Anticoagulation with Focus on Atrial Fibrillation. PLoS One. 2015 May 22;10(5):e0124719. doi: 10.1371/journal.pone.0124719. eCollection 2015. PMID 26001109